Protocol Title: Evaluating the addition of obturator nerve block to adductor canal block for total knee arthroplasty

Statistical Analysis Plan

PI: Christina Jeng

NCT03326999

Date: Sept 29, 2017

Prior to the beginning of the study, a sample size calculation was performed and was based on an  $\alpha$  of 0.05 and a  $\beta$  of 0.2. Patients were randomized into an intervention and control group. Baseline characteristics of subjects in each group were compared using chi-square tests for categorical variables and independent t-tests for continuous variables. No significant differences were detected between the baseline characteristics of each group; thus, direct comparisons of the outcomes of each group were analyzed. For categorical variables, chi-square tests were utilized, unless one value in the 2x2 matrix was under 5, in which case Fischer's exact test was utilized. For binary tests, odds ratios with 95% confidence intervals were reported. For continuous variables, independent t-test was used. All calculations were performed via SAS Statistical Software (Cary, NC).